CLINICAL TRIAL: NCT05590663
Title: Functional Activity Scoring Tool (FAST) and Patient-Specific Functional Scale (PSFS): Assessment and Validation of Two Functional Scales in Patients With Knee Osteoarthritis (OA) in Singapore
Brief Title: FAST and PSFS: Assessment and Validation of Two Functional Scales in Patients With Knee OA in Singapore
Status: Completed | Type: Observational
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Singapore Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 202206-00049
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee injury and Osteoarthritis Outcome Score; Patient-Specific Functional Scale; Functional Activity Scoring Tool; Functional assessment
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis: Individuals who are medically diagnosed with knee osteoarthritis and eligible for physiotherapy care in SingHealth Polyclinics will be recruited. Inclusion criteria include: individuals above the age of 45, proficient in colloquial/conversational English, and diagnosed with knee osteoarthritis. Exclusion criteria include additional underlying medical or trauma conditions of the knees (e.g., trauma, fracture, infection, inflammatory disease, tumour), history of knee surgery within the last three months, or clinically recognizable cognitive impairment that inhibits the completion of the questionnaires.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — routine referral-based physiotherapy treatment for patients with knee osteoarthritis

SUMMARY:
The new National One-Rehab framework mandates the use of the Patient-Specific Functional Scale (PSFS) as an outcome measure to track patients' rehabilitation progress. Anecdotally, we have encountered patients (especially elderly ≥ 65 years old) with difficulty understanding and completing such questionnaire accurately. We developed a pictorial functional scale (Functional Activity Scoring Tool, FAST) with reference to the successful application of the Wong-Baker FACES pain rating scale. Concurrently, we hope to validate PSFS and FAST against Knee injury and Osteoarthritis Outcome Score (KOOS) which is validated in Singapore population.

This study aims to investigate the reliability and validity of the PSFS and FAST in patients with knee osteoarthritis. We hypothesize that both the PSFS and FAST can be used to measure difficulty in performing activities of daily living in patients with knee osteoarthritis in a reliable and valid manner.

The FAST and PSFS questionnaires will be administered to patients in SingHealth Polyclinics with knee osteoarthritis to explore the psychometric and clinimetric properties. Eligibility criteria were: age 45 and above, proficient in English, diagnosed with knee osteoarthritis. Patients were excluded if they have underlying medical or trauma conditions (i.e., trauma, fracture, infection, inflammatory disease, tumor), history of knee surgery within the last 3 months, or clinically recognizable cognitive impairment.

Eligible patients will be informed about the purpose of the study and the confidentiality and anonymity of the process. After giving written consent they will complete a questionnaire on demographic and clinical characteristics and the sets of outcome measures (FAST, KOOS, PSFS). Participants will then return at two-to-three weeks later to complete the sets of outcome measures again and GROC, and to state their preferred outcome measures. Statistical analysis will be conducted to evaluate the validity and reliability of PSFS and FAST against KOOS.

DETAILED DESCRIPTION:
Validation

The FAST and PSFS questionnaires will be administered to patients in SingHealth Polyclinics (SHP) with knee osteoarthritis to explore the psychometric and clinimetric properties. Eligibility criteria were: age 45 and above, proficient in English, diagnosed with knee osteoarthritis. Patients were excluded if they have underlying medical or trauma conditions (i.e., trauma, fracture, infection, inflammatory disease, tumor), history of knee surgery within the last 3 months, or clinically recognizable cognitive impairment. Statistical analysis will be conducted to evaluate the validity and reliability of PSFS and FAST against KOOS.

Questionnaire

1. FAST

   FAST is developed by Mr. Tang Zhi Yin and Mr. Ng Khim Siong from SHP physiotherapy department. It is a pictorial scale with 7 emotion faces (different degrees of sadness to happiness) on stairs to depict corresponding level of difficulty a patient is experiencing during performing activity. Short descriptions are labelled under the faces, as well as a scale of 0-10 to guide the patient to rate his/her functional difficulty. The patient is asked to identify up to 3 activities that being affected due to his/her current musculoskeletal pain, and to rate each activity on the FAST.
2. PSFS

   The PSFS is a self-reported, patient-specific measure that assesses patients' functional status. Patients are asked to identify three activities that are most affected by their condition and then rate their ability on a 0-10 scale, where 0 is unable to perform activity and 10 is able to perform activity at the same level as before the onset of symptoms.
3. KOOS

   The KOOS is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. It is a validated tool in Singapore for knee osteoarthritis patients. It has a total of 42 items in 5 subscales i.e., pain, other symptoms, function in daily living, function in sport and recreation, and knee-related quality of life. Scores are interpreted independently for each subscale. As our study focuses on function, we only apply subscales for function in daily living, function in sport and recreation, and knee-related quality of life.
4. GROC

The GROC is an outcome measure that assesses patients' self-perception of change in their condition between sessions. Participants were asked to rate the change in their condition on a 15-point transitional scale from -7 (a very great deal worse) to 7 (a very great deal better). The GROC scale is easy to administer, requires minimal skills or training, has good reproducibility, and is sensitive to change.

Data collection

Eligible patients will be informed for the purpose of the study and the confidentiality and anonymity of the process. After giving written consent they will complete a questionnaire on demographic and clinical characteristics and the sets of outcome measures (FAST, KOOS, PSFS). Participants will then return at two-to-three weeks later to complete the sets of outcome measures again and GROC, and to state their preferred outcome measures.

Statistical analysis

All statistical analysis will be conducted using SPSS 26 for Windows. To investigate validity, the discriminant validity was evaluated by the Spearman correlation coefficient according to the following criteria: high (rho ≥ 0.60); moderate (rho < 0.60 - ≥ 0.30); or low (rho <0.30). To analyze the test-retest reliability, the intraclass correlation coefficient (ICC) is calculated. An ICC value of less than 0.40 indicated poor reliability, whereas values between 0.40 and 0.75 indicated fair to good reliability; an ICC value of greater than 0.75 showed excellent reliability.

ELIGIBILITY:
Inclusion criteria:

* individuals above the age of 45
* proficient in colloquial/conversational English
* diagnosed with knee osteoarthritis.

Exclusion criteria:

* additional underlying medical or trauma conditions of the knees (e.g., trauma, fracture, infection, inflammatory disease, tumour)
* history of knee surgery within the last three months
* clinically recognizable cognitive impairment that inhibits the completion of the questionnaires.

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in functional status as assessed by Functional Activity Scoring Tool (FAST) | 3 weeks from baseline examination
  Change in functional status as assessed by FAST using a points system
Change in functional status as assessed by Patient-Specific Functional Scale (PSFS) | 3 weeks from baseline examination
  Change in functional status as assessed by PSFS using a points system
Change in functional status as assessed by Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 weeks from baseline examination
  Change in functional status as assessed by KOOS using a points system
Patients' self-perception of change in their knee condition as assessed by Global Rating of Change Score (GROC) | 3 weeks from baseline examination
  Patients' self-perception of change in their knee condition as assessed by GROC using a points system

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yin Tang, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that will be shared include:
  * Demographics data
  * Outcome data for primary and secondary endpoints
Time Frame: IPD will be available beginning 6 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Data will be made available to qualified researchers upon reasonable request, subject to approval by the sponsor and completion of a data use agreement.

REFERENCES:
- [Background] Stratford P, Gill C, Westaway M, Binkley J. Assessing disability and change on individual patients: a report of a patient specific measure. Physiotherapy Canada. 1995;47(4):258-63.
- [Background] Chatman AB, Hyams SP, Neel JM, Binkley JM, Stratford PW, Schomberg A, Stabler M. The Patient-Specific Functional Scale: measurement properties in patients with knee dysfunction. Phys Ther. 1997 Aug;77(8):820-9. doi: 10.1093/ptj/77.8.820. PMID 9256870
- [Background] Xie F, Li SC, Roos EM, Fong KY, Lo NN, Yeo SJ, Yang KY, Yeo W, Chong HC, Thumboo J. Cross-cultural adaptation and validation of Singapore English and Chinese versions of the Knee injury and Osteoarthritis Outcome Score (KOOS) in Asians with knee osteoarthritis in Singapore. Osteoarthritis Cartilage. 2006 Nov;14(11):1098-103. doi: 10.1016/j.joca.2006.05.005. Epub 2006 Jun 30. PMID 16814575
- [Derived] Tang ZY, Ng KS, Tee JX, Lee EZE, Bistamam MHB, Wong JS, Koh YLE, Yeung M. Validation of the Functional Activity Scoring Tool (FAST): a novel pictorial scale for assessing function in patients with knee osteoarthritis in primary care. BMJ Open. 2025 Aug 31;15(8):e100732. doi: 10.1136/bmjopen-2025-100732. PMID 40887119
- [Derived] Tang ZY, Ng KS, Koh YLE, Yeung MT. Study protocol for the validation of a new pictorial functional scale in patients with knee osteoarthritis: the functional activity scoring tool (FAST). BMJ Open. 2024 Jan 8;14(1):e076947. doi: 10.1136/bmjopen-2023-076947. PMID 38191249